CLINICAL TRIAL: NCT07081048
Title: THE EFFECT OF BUZZY® AND SHOTBLOKER® APPLICATION ON THE PAIN AND COMFORT LEVEL OF NEWBORNS DURING HEEL PRICK BLOOD SAMPLING IN NEWBORNS
Brief Title: Pain and Comfort Levels During Heel Stick Blood Sampling in Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Duygu Sonmez Duzkaya, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025/03
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Newborn
Keywords: pain; confort; Buzzy; Shotbloker
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy® Group (Experimental): The ice pack, which has been removed from the deep freezer in advance, should be left at room temperature for 10 minutes, and the hole in the ice pack should be placed on the hook behind the Buzzy®. Buzzy® will be placed on the lateral side of the left heel and activated for 30 seconds. After 30 seconds, Buzzy® will be pulled up 1 centimetre (cm), and the heel will be punctured with a sterile lancet to collect blood on the Guthrie card. After the heel blood collection procedure, Buzzy® will be pulled back to the punctured heel area and left for another 30 seconds.
  Interventions: Other: Buzzy®.Group
- Shotbloker® Group (Experimental): ShotBlocker will be placed on the designated area for collecting the baby's heel blood. After ensuring that the protrusions of the ShotBlocker are in contact, pressure will be applied for 20 seconds.
  The heel will be punctured with a sterile lancet in the area designed for applying the ShotBlocker, and the ShotBlocker will be removed from the area. The blood collected will be collected on Guthrie paper.
  Interventions: Other: ShotBlocker Group
- Control Group (No Intervention): Without any intervention or application to the heel area, the lateral side of the left foot will be punctured with a lancet of the same type, and heel blood sampling will be performed according to the clinic's routine practice. At the clinic, heel blood sampling is performed without any intervention, with the baby in the mother's arms.

INTERVENTIONS:
Other: Buzzy®.Group — The ice pack, which has been removed from the deep freezer in advance, should be left at room temperature for 10 minutes, and the hole in the ice pack should be placed on the hook behind the Buzzy® will be placed on the lateral side of the left heel and activated for 30 seconds. After 30 seconds, Buzzy® will be pulled up 1 centimetre (cm), and the heel will be punctured with a sterile lancet to collect blood on the Guthrie card. After the heel blood collection procedure, Buzzy® will be pulled back to the punctured heel area and left for another 30 seconds.
  Arms: Buzzy® Group
Other: ShotBlocker Group — ShotBlocker will be placed on the designated area for collecting the baby's heel blood. After ensuring that the protrusions of the ShotBlocker are in contact, pressure will be applied for 20 seconds.
  The heel will be punctured with a sterile lancet in the area designed for applying the ShotBlocker, and the ShotBlocker will be removed from the area. The blood collected will be collected on Guthrie paper.
  Arms: Shotbloker® Group

SUMMARY:
Aim: The study was designed to determine the effect of Buzzy® and Shotbloker® application on pain and comfort levels in newborns during heel pricking. Method:The study was a randomised controlled trial. The study sample consisted of 159 newborns (Buzzy: 53, Shotbloker: 53, control: 53) who had heel pricks between March 2025 and December 2025 at the Samandağ State Hospital Neonatal Care Unit. The data collection tools used will be the Newborn Information Form, the Newborn Pain Scale, the Newborn Comfort Behaviour Scale, and the Buzzy® and Shotbloker® devices. In the intervention group, the Buzzy® and Shotbloker® devices will be applied before and after heel pricking, while the control group will receive routine care. The infants' pain and comfort levels will be assessed by the nurse before and after the procedure.

DETAILED DESCRIPTION:
The study was designed as a randomised controlled trial to determine the effect of Buzzy® and Shotbloker® application on pain and comfort levels in newborns during heel prick blood sampling.

Materials and Methods Setting After obtaining ethical committee approval, the study will be conducted with babies admitted to the Neonatal Unit of Samandağ State Hospital between March and December 2025.

Sample According to the power analysis performed for the sample size, the power of the sample was calculated using the G*Power 3.1 programme in line with the literature. With a Type I error rate of 0.05 and a test power of 0.80 (α = 0.05, 1-β = 0.80), the minimum sample size (with 53 newborns in each group) was calculated to be 159.

Data Collection In the study, babies brought to the Neonatal Unit for heel prick blood sampling will first be evaluated according to the sampling criteria, and those who do not meet the criteria will be excluded from the study. The nurse researcher herself will collect the data, evaluate it using the NIPS pain scale and the Neonatal Comfort Behaviour Scale, collect the heel blood, and administer the Buzzy® and Shotbloker® applications. To ensure consistency in the application, heel blood will be collected from the left lateral foot of all infants included in the study by the same nurse.

Application Before the heel prick procedure, the room will be well lit and warm to ensure that the babies are comfortable. Babies in the Buzzy, Shotbloker, and control groups who meet the sample criteria will first be examined by a paediatrician, and if there are no contraindications for heel pricking, their parents will be informed about the study and their verbal and written consent will be obtained, after which the data collection form will be completed. The 'Baby Information Form' will be completed by the researcher before the heel pricking procedure. Immediately afterwards, the infant's physiological parameters (pulse, SpO2) will be measured, and the infant's pain and comfort will be assessed by the researcher using the NIPS Scale and YDKÖ. All infants participating in the study will be held in their mothers' arms during the heel prick procedure.

Before taking blood, the nurse will clean the skin with 70% isopropyl alcohol and wait for it to dry. Blood will be taken from each baby using a single sterile lancet, and the first drop of blood will be wiped away. Then, a blood sample will be taken from one side of the Guthrie card, covering the entire marked area. The blood sample will be taken so that bloodstains of equal size are visible on both sides of the blood collection paper. In this way, each of the five marked areas will be filled. During blood collection, the blood collection paper will not be pressed, and the heel will not be squeezed excessively to prevent haemolysis or dilution (thinning) of the blood with tissue fluid. All heel blood samples will be collected on standard blood sample paper containing five circles. After heel blood collection, the researcher will measure the physiological parameters of the babies in the Buzzy group, Shotbloker group, or control group a second time and record their pain and comfort assessments.

STATISTICAL ANALYSIS The data obtained within the scope of the research will be evaluated using the Statistical Package For Social Science (SPSS) 22.0 software package. The Chi-square Fisher's exact test will be used to determine the homogeneity between groups, the Independent Groups t-test will be used to determine whether the difference between groups is statistically significant, and the One-Way Analysis of Variance will be used to determine which group the difference originates from using the Bonferroni test.

One-Way Analysis of Variance will be used to determine whether the difference is statistically significant between groups, and the Bonferroni test will be used to determine which group the difference originates from. A significance level of 0.05 will be used, and if p<0.05, a significant difference will be determined, and if p>0.05, no significant difference will be determined.

ELIGIBILITY:
Inclusion Criteria:

* The baby must be full-term (38-42 weeks),
* No analgesic administration up to 8 hours prior to the procedure,
* No pain prior to the procedure,
* No chronic or metabolic disease,
* Born at least 24 hours prior,
* Being in the hospital during the study period

Exclusion Criteria:

* The baby is not full-term,
* Analgesic medication has been administered within 8 hours prior to the procedure,
* The baby has a chronic or metabolic disease,
* The baby requires oxygen support,
* The baby cannot be fed orally,
* The baby is not in the hospital on the dates the study will be conducted and the parents do not agree to participate in the study.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 1 day
  The Neonatal Infant Pain Scale (NIPS) was developed by Lawrence and colleagues in 1993. Its validity and reliability in Turkish were established by Akdovan in 1999 (81). Reliability values were found to be 0.83, 0.83, and 0.86 before, during, and after the procedure, respectively. The neonatal infant pain scale assesses facial expressions (0; relaxed, 1; distressed), crying (0; no crying, 1; whimpering, 2; loud crying), breathing (0; relaxed, 1; variable-irregular), arm (0; relaxed-free, 1; flexion-extension), legs (0; relaxed-free, 1; flexion-extension), and sleep-wakefulness (0; sleeping-awake and calm, 1; restless). Pain is assessed based on the total score. After observation, the scale is scored from a maximum of 7 to a minimum of 0. According to the scale, a score of 7 indicates the highest level of pain, while a score of 0 indicates the lowest level of pain. If the NIPS score is between 0 and 2, the pain is considered to be absent or mild. If the pain score is between 3 and 4, i
Newborn Information Form | 1 day
  The information form has been prepared by reviewing the relevant literature and includes the baby's gestational age, gender, birth weight, birth length, mode of delivery, pre- and post-procedure physiological parameters (SPO2, pulse), NIPS Pain Score, and Newborn Comfort Behaviour Scale. The data collection form contains a total of 6 questions.
Newborn Comfort Behaviour Scale (NCBS) | 1 day
  The scale was first developed in 1992 by Ambuel and colleagues to assess distress in patients receiving mechanical ventilator support in a paediatric intensive care unit. Later, in 2009, Van Dijk and colleagues revised the scale and established the validity and reliability of the COMFORTneo scale for measuring behaviour in newborns without physiological parameters.
  The COMFORTneo scale (NCBS) consists of 6 parameters (alertness, calmness/agitation, The COMFORTneo scale (YKDÖ) is a Likert-type scale consisting of six parameters (alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, muscle tone). It is also a tool that provides nurses with numerical data to assess the comfort of newborns. The scale was revised in 2014 by Karaman et al. to establish its 'Turkish Validity and Reliability.' The lowest score on the scale is 6 and the highest score is 30, with high scores indicating that the baby is not comfortable. The Cronbach's alpha coefficient of t

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] • Inal, S., Aydin Yilmaz, D., & Erdim, L. (2022). The effectiveness of swaddling and maternal holding applied during heel blood collection on pain level of healthy term newborns; randomized controlled trial. Early Child Development and Care, 192(13), 2066-2077.
- [Background] Yavas S, Bulbul T, Topcu Gavas H. The effect on pain level and comfort of foot massages given by mothers to newborns before heel lancing: Double-blind randomized controlled study. Jpn J Nurs Sci. 2021 Oct;18(4):e12421. doi: 10.1111/jjns.12421. Epub 2021 Apr 20. PMID 33880884
- [Background] van der Burg S, Oerlemans A. Fostering caring relationships: Suggestions to rethink liberal perspectives on the ethics of newborn screening. Bioethics. 2018 Mar;32(3):171-183. doi: 10.1111/bioe.12425. PMID 29442381
- [Background] Sok P, Lupo PJ, Richard MA, Rabin KR, Ehli EA, Kallsen NA, Davies GE, Scheurer ME, Brown AL. Utilization of archived neonatal dried blood spots for genome-wide genotyping. PLoS One. 2020 Feb 21;15(2):e0229352. doi: 10.1371/journal.pone.0229352. eCollection 2020. PMID 32084225
- [Background] Shah SR, Kadage S, Sinn J. Trial of Music, Sucrose, and Combination Therapy for Pain Relief during Heel Prick Procedures in Neonates. J Pediatr. 2017 Nov;190:153-158.e2. doi: 10.1016/j.jpeds.2017.08.003. PMID 29144240
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830
- [Background] Anand KJ, Hickey PR. Pain and its effects in the human neonate and fetus. N Engl J Med. 1987 Nov 19;317(21):1321-9. doi: 10.1056/NEJM198711193172105. No abstract available. PMID 3317037